CLINICAL TRIAL: NCT04069832
Title: Evaluating the Single-Session Consultation Service at the Krasner Psychological Center and Putnam
Acronym: SSC@KPC&Putnam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Jessica Schleider, Assistant Professor of Psychology, Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB2019-00362
Record Dates: First submitted 2019-08-21; First posted 2019-08-28 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Mental Health Impairment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): SINGLE-SESSION CONSULTATION
  Interventions: Behavioral: Single-Session Consultation

INTERVENTIONS:
Behavioral: Single-Session Consultation — A single, goal-directed consultation session based on Solution-Focused Brief Therapy (SFBT). SFBT is an evidence-based therapy approach that is primarily focused on the client's present problems and their immediate future. When using SFBT in a single-session the aim of the intervention becomes empowering the client to take the smallest possible steps towards their desired future.
  Other Names: SSC

SUMMARY:
Stony Brook University is home to several mental health clinics, that all work towards achieving overall wellness of their clients. The goals of Stony Brook University are met with the help of associated clinics that strive to improve wellness of individuals and their communities by helping to treat both mental and physical health impairments. Two of these many clinics are the Krasner Psychological Center (KPC), and the Mind Body Clinical Research Center (MBCRC)..

At present, the KPC and MBCRC face a challenge common to virtually all mental health clinics across the United States: the demand for psychological services far outpaces the number of available providers. Indeed, in the US, approximately 70% of those in need of mental health services do not receive them. As such, wait-lists at mental health clinics like the KPC and MBCRC are increasingly long, and longer wait-times for psychotherapy have predicted worse clinical outcomes once treatment is accessed (i.e., a 'nocebo' effect). Thus, there is a pressing need for effective, sustainable service delivery models that may facilitate more rapid access to care-for instance, providing a low-intensity service rapidly after an individual decides to seek treatment, capitalizing on client motivation. This sort of rapidly-provided, low-intensity service might have the added benefit of reducing overall waitlist lengths--e.g., if some subset of clients find the low-intensity service to be sufficient, a single session might be sufficient (in some cases) to spur positive behavioral and emotional change.

One solution to this problem is the integration of single-session services into mental health clinics. Extensive research suggests that both youths and adults can benefit from just one session of goal-directed counseling, and these clinical benefits have been observed for a wide array of problems-including anxiety, depression, self-harm, and interpersonal conflicts. This research suggests the possibility that, for some subset of clients, a single session of counseling may be helpful, or even sufficient, in reducing clinical distress. Therefore, the objective of this study is to examine the feasibility, acceptability, and short-term effects of the new Single-Session Consultation (SSC) service, which is presently being provided to clients on the waiting list for psychotherapeutic services at the Krasner Psychological Center and the Mind Body Clinical Research Center. The SSC offers clients the opportunity to participate in a single, goal-directed consultation session based on Solution-Focused Brief Therapy (SFBT) within two weeks of inquiring about services at the KPC and MBCRC (typically, clients wait 2-6 months prior to their initial clinic appointment). SFBT is an evidence-based therapy approach that guides services offered by existing single-session therapy clinics internationally. Clients who participate in the SSC at any of these clinics may find the session helpful; two weeks after participating in the session, they receive the option to remain on the waitlist for long-term psychotherapy or remove themselves from the waitlist for psychotherapy, depending on whether they feel their clinical needs have been successfully addressed.

DETAILED DESCRIPTION:
The Stony Brook University (SBU) clinical psychology doctoral program is currently ranked 4th among the top clinical psychology doctoral programs in the country (2016, U.S. News and World Report, Best Graduate Schools) and is accredited by both the APA Committee on Accreditation (APA CoA) and the Psychological Clinical Science Accreditation System (PCSAS). The Krasner Psychological Center (KPC) is a psychology training clinic housed in the Department of Psychology and associated with the doctoral program in clinical psychology at SBU. The mission of the KPC is twofold, namely, (a) to provide high quality experiential training in the delivery of psychological services to trainees in the associated 3 doctoral program, as well as to externs, doctoral interns, and post-doctoral residents; and (b) to provide evidence-based mental health services to the nearby communities. All supervisors at the KPC are doctoral-level psychologists. Psychotherapy services at the KPC are based on Cognitive-Behavior Therapy models and include weekly, outpatient psychotherapy for a wide range of problems in children and adults; therapy is designed to be short-term, personalized, and effective in empowering clients to manage their symptoms and distress.

Similarly, the Mind Body Clinical Research Center (MBCRC) bases their interventions on evidence-based practices that address multiple factors associated with health impairments. Additionally, they focus on providing comprehensive psychiatric evaluations and assessments to aid in the creation of adequate treatment plans. The MBCRC specifically focuses on using mind-body to help identify risk and resiliency factors associated with mental health outcomes in their clients. This technique works in support of the scientific link that has been shown to exist between our mental/physical health with overall wellness and quality of life. Using this technique, the MBCRC is able to help individuals make changes early on that can help to prevent worsening symptomology of mental illness, preserve physical health, and make improvements in overall wellness.

The single-session consultation, a one-time service provided to adolescents and adults on the clinics' waitlist (which may extend from 2 to 6 months), includes components of Solution-Focused Brief Therapy (SFBT). SFBT lends itself naturally to the single-session format in that it focuses on the present and future, targeting the desired outcome of therapy, a future in which the primary problem is absent or less influential. Importantly, SFBT providers focus on the factors that maintain/underlie solutions rather than the factors than maintain/underlie problems.

GENERAL SCREENING PROCEDURES

When individuals seeking services at the KPC and MBCRC express interest in scheduling an appointment with a clinician, they are first instructed (by phone) about the clinical and research aims by the clinic's clinical research coordinator. The clinical research coordinator is a trained, independent staff member and is not involved in the provision of psychotherapy or single-session consultation services. The clinical research coordinator conducts a standardized, structured phone screen with the individual to identify primary reasons for seeking mental health services and to assess the appropriateness of presenting concerns for treatment at the KPC or MBCRC. If the individual is eligible to receive services at one of our clinics (i.e., if their concerns fall within the scope of clinical problems treated; if the individual/family is English-speaking; and if problems are not so acute as to require immediate hospitalization, in which case they are referred to the nearest emergency room), the client is placed on the waitlist for psychotherapy services.

During the same phone call, if the identified patient is 13 years or older, the clinical research coordinator then introduces the opportunity to participate in the Single Session Consultation (SSC) service at the KPC or MBCRC.

The clinical research coordinator indicates that as part of SSC service participation the client will be asked to complete questionnaires in order to provide their clinician with information about their current mental health, and for the purposes of planning and assessing the usefulness of services. The clinical research coordinator will also indicate that the individual may opt to allow or not allow us to use this data for research purposes. They will be informed that if they do choose to allow their data to be used for research, it will be de-identified and combined with other patient data for the purposes of understanding how well our treatment programs work for different types of individuals. The coordinator will emphasize that their choice to participate, or not participate in research will NOT impact their eligibility for the SSC service or longer-term psychotherapy in any way.

The clinical research coordinator will again review the purpose of the research study and obtain fully informed consent at the beginning of the patient's in-person intake visit. A private clinic room will be available for this purpose. Adult patients (or adolescent patient and her/his parent) can either agree or disagree to allow the research team to use their clinical data for research by checking the appropriate check-box on the paper consent form. Patients will also be able to elect to participate in the specific study described in the consent form and/or to have their de-identified data added to a registry for future unspecified research projects. Obtaining consent verbally by phone and in person at the initial intake visit will allow patients to ask questions and minimize the risk of coercion.

DATA COLLECTION PROCEDURES SPECIFIC TO THE SINGLE-SESSION CONSULTATION SERVICE

The following measures will be administered to clients immediately prior to participation in the SSC:

* Brief Personal Data Questionnaire (Adult or Adolescent version)
* State Hope Scale (assessing 'agency')
* Brief Hopelessness Scale (assessing 'hope/hopelessness')
* Brief Symptom Inventory - 18

Then, immediately following the one-hour SSC session, participants will be asked to complete immediate post-SSC questionnaires:

* State Hope Scale (assessing 'agency')
* Brief Hopelessness Scale (assessing 'hope/hopelessness')
* Consultation Feedback Form

Finally, two weeks after completing the SSC, the clinical research coordinator will contact the client via phone to administer the Brief Symptom Inventory a second time. At the end of this phone call, the clinical research coordinator will then give the client the option to remain on the waitlist for long-term psychotherapy or remove themselves from the waitlist for psychotherapy, depending on whether they feel their clinical needs have been successfully addressed.

For therapists, "Therapist beliefs about SSC" measure will be administered before SSC training, immediately after SSC training, and two months after the SSC training date.

NOTE 1: A client may reschedule an SSC session if they are unable to attend it. The KPC and MBCRC will not limit the number of times a client is permitted to reschedule an SSC session, should they remain interested in receiving one. Additionally, if clients endorse significant clinical risk (to themselves or others) while participating in the study, study procedures may be interrupted (e.g., an SSC session may be terminated in order to address urgent clinical needs). If a client's initial SSC session is interrupted or terminated due to a need to address urgent clinical risk, the client will be permitted to reschedule their SSC session for a later date.

NOTE 2: If a participant does not respond to the clinic's requests for a 2-week follow-up phone call within two weeks of being contacted, per KPC and MBCRC policy, it will be assumed that the client is no longer interested in services and will be removed from the waiting list. Pre-to-post SSC data for these clients will still be used for analyses unless they request that their data not be used in the study.

NOTE 3: The lead investigator (Jessica Schleider) will train all SSC clinicians prior to their delivering SSC sessions with clients. This training will be approximately 2 hours in length and will review the principles and key elements of the SSC protocol, in addition to challenges that might emerge while delivering the SSC. The written SSC protocol used by clinicians in the study will be made publicly available by the Principal Investigator upon project completion.

ELIGIBILITY:
Inclusion Criteria:

* All adolescent (ages 13+) and adult clients on the waitlist for clinical psychotherapy services at the KPC and MBCRC will be eligible to take part in this research.

Exclusion Criteria:

* Child clients at the KPC and MBCRC under the age of 13 will not be eligible to participate in this study, because the Single-Session Consultation service presently being offered at the KPC and MBCRC is designed for use with adolescents and adults (i.e., it would be developmentally inappropriate for younger children.).
* Non-English speaking individuals will not be eligible to receive any clinical services at the KPC and MBCRC because all therapists at the clinics are English-speaking.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Change in State Hope Scale score ('agency') | Pre-Single-Session Consultation (SSC) & immediately Post-SSC (1-3 minutes post-intervention))
  The State Hope Scale is a 6 item self-report measure of agentic, goal-directed thinking. Respondents rate 6 items on a Likert scale from 1 (definitely false) to 8 (definitely true). Higher mean scores reflect a greater sense of personal agency (i.e., personal capacity to pursue and sense of having attained goals). Scores range from 1-8.
Change in Beck Hopelessness Scale - 4 item version score ('hope') | Pre-Single-Session Consultation (SSC) & immediately Post-SSC (1-3 minutes post-intervention))
  Respondents report agreement with 4 items, each rated on a 0-3 scale, indicating levels of hopelessness about the future. Higher summed scores reflect greater levels of hopelessness, and scores range from 0-12.

SECONDARY OUTCOMES:
Change in Brief Symptom Inventory-18 | Pre-SSC & 2 week follow-up
  The Brief Symptom Inventory-18 (BSI-18) assesses self reported psychopathology and distress. Respondents rate endorsement of 18 physical and emotional complaints on a 0-4 Likert scale. The total sum score yields an additional total distress score (range: 0-72). Higher scores indicate higher levels of overall psychological distress.
Consultation Feedback Form | Immediately Post-SSC (1-3 minutes post-intervention) only
  The consultation feedback form contains 5 items, rated on a 1 ("Not at all") to 5 ("Very much") Likert scale, indicating endorsement of a series of statements about responses to the Single Session Consultation program (e.g., "Did you find the consultation helpful in addressing your concern(s)?" and "How hopeful are you that the action plan will be useful?." Higher mean scores across these 5 items indicates greater perceived usefulness of the SSC.
Therapist Beliefs about SSC | Pre-SSC Training, Immediately post-SSC training, and 2 months after SSC training
  A brief measure examining therapists' perceived acceptability, feasibility, and effectiveness of the Single Session Consultation (SSC) program. The measure is comprised of questions rated on a 1 ("Completely Disagree") to 5 ("Completely Agree") scale, indicating endorsement of a series of statements about the Single Session Consultation Program, and short answer questions. Higher mean scores across these 5 items indicate greater perceived acceptability, feasibility, and effectiveness of the SSC. This measure will be administered to clinicians at Mind Body Research Center and Adolescent Outpatient Psychiatry only due to the delayed addition of this measure.

OTHER OUTCOMES:
Brief Personal Data Questionnaire (Adult or Adolescent version) | Pre-SSC only
  On this survey, participants report basic demographic information; whether they have a history of receiving past psychotherapy; whether they have a history of receiving past medication; and complete qualitative, open-ended questions on the nature of their presenting problem (i.e., why they have chosen to seek treatment). Because this is a demographic questionnaire, no scores are associated with this measure.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L Schleider, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data will be made available on Open Science Framework upon conclusion of the pilot study (N= 60).
Supporting Information: Study Protocol, SAP, ICF

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-02-13): https://cdn.clinicaltrials.gov/large-docs/32/NCT04069832/SAP_002.pdf